CLINICAL TRIAL: NCT01666626
Title: Investigating Ultrasound Stiffness Imaging for Predicting Outcomes in Crohn's Disease
Brief Title: Ultrasound Stiffness Imaging in Crohn's Disease
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: Crohn's and Colitis Foundation (Other)
Responsible Party: Principal Investigator, Ryan W. Stidham, Principle Investigator, University of Michigan
Other Study IDs: HUM64431
Record Dates: First submitted 2012-08-07; First posted 2012-08-16 (Estimated); Last update posted 2015-07-30 (Estimated); Status verified 2015-07

CONDITIONS: Crohn's Disease; Ultrasound; Intestinal Fibrosis; Shear Wave Imaging; Acoustic Radiation Force Impulse
Keywords: crohn's disease; ultrasound; intestinal fibrosis; shear wave imaging; acoustic radiation force impulse
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Crohn's Inpatients: Crohn's Inpatients, with clinical small bowel obstruction All undergo ultrasound stiffness imaging (USI) of distal affected ileum.
  Interventions: Procedure: Ultrasound stiffness imaging
- Crohn's Outpatients: Crohn's Outpatients, starting anti-TNF therapy All undergo ultrasound stiffness imaging (USI) at week 0, 6, 14
  Interventions: Procedure: Ultrasound stiffness imaging

INTERVENTIONS:
Procedure: Ultrasound stiffness imaging — Subjects will undergo transabdominal ultrasound of the distal intestine. Distal intestine motion capture will be used for off-line stiffness assessment by two-dimensional speckle tracking. In addition, shear wave imaging will be used for real-time stiffness assessment.

SUMMARY:
The purpose of this study is to determine whether ultrasound-based assessment of intestinal stiffness in patients with Crohn's disease predicts the effectiveness of medical therapy or the need for surgical resection.

DETAILED DESCRIPTION:
Modern medical therapy in Crohn's disease, including immunomodulators and biologic compounds, has revolutionized disease treatment. However, a significant portion of individuals will not respond to medications, most often due to the development of intestinal fibrosis. Over the course of Crohn's disease repeated episodes of inflammation and abnormal wound healing lead to progressive intestinal fibrosis, strictures, and bowel obstruction. While inflammatory Crohn's disease often responds to medical therapy, predominantly fibrostenotic intestinal disease is unresponsive and requires surgery. Our inability to accurately distinguish intestinal inflammation from fibrosis frequently leads to empiric trials of steroids and immunosuppressive therapies. This often proves futile, delays inevitable surgery, and unnecessarily exposes the patient to medication-related risks for months and sometimes years. At present there are no available means to distinguish medically responsive inflammatory disease from predominately fibrotic intestinal disease. The unmet need in this field is an accurate diagnostic technology to determine which patients will benefit from anti-inflammatory therapy, and which patients should go directly to surgery. Non-invasive ultrasound stiffness imaging (USI) may be a surrogate marker of underlying bowel wall fibrosis that aids in predicting if Crohn's disease will be responsive to medical therapy.

Two USI methods have recently been developed: Ultrasound elasticity imaging (UEI) uses 2D speckle-tracking to measure tissue strain, a surrogate of fibrosis. The second, shear wave imaging (SWI), is a commercially available technology that measures the speed of ultrasonic shear waves through tissue. Shear waves travel more rapidly through stiff tissue. The central hypothesis of this proposal is that ultrasound stiffness imaging (USI) quantitatively distinguishes predominately inflammatory from fibrotic bowel wall thickening, and therefore is predictive of the likelihood of response to medical therapy or the need for surgery.

We plan to objectively test our central hypothesis and attain the objective of this application by pursuing the following three specific aims:

Specific Aim 1 (SA-1): Determine if USI stiffness measurements of intestinal strictures in Crohn's patients admitted with small bowel obstruction predicts response or failure of medical therapy based on CDAI and objective inflammatory biomarkers during index hospitalization and at 90 day follow-up.

Inpatient Inclusion Criteria:

* Subjects must be 18 years of age or older
* Previous diagnosis of Crohn's disease with imaging demonstrating involvement of the ileum
* Hospital admission imaging demonstrating small bowel dilation (to > 3.5 cm)
* CDAI score of >220.

Inpatient Exclusion Criteria:

* Active Clostridium difficile colitis/enteritis
* Presence of abdominal enterocutaneous fistulas in the ultrasound path.
* Prior abdominal hernia repair with mesh placement in the ultrasound path.

Specific Aim 2 (SA-2): Determine if USI stiffness measurements of diseased ileum in Crohn's outpatients starting Anti-Tumor Necrosis Factor-Alpha therapy predicts response to medical therapy based on CDAI and objective inflammatory biomarkers.

Outpatient Inclusion Criteria

* Crohn's patients age 18 and over starting anti-TNF therapy
* CDAI score > 220 to denote clinical disease activity.

Outpatient Exclusion Criteria:

* Active Clostridium difficile colitis/enteritis
* Presence of abdominal enterocutaneous fistulas in the ultrasound path
* Prior abdominal hernia repair with mesh placement in the ultrasound path
* Current use of prednisone or budesonide
* Changing anti-TNF due to allergy (including a TNF-induced lupus-like arthritis).

ELIGIBILITY:
Inclusion Criteria:

* CDAI score >220
* if INPATIENT: admission for small bowel obstruction.
* if OUTPATIENT: start of anti-tumor necrosis alpha therapy

Exclusion Criteria:

* Active Clostridium difficile colitis/enteritis
* Presence of abdominal enterocutaneous fistulas in the ultrasound path
* Prior abdominal hernia repair with mesh placement in the ultrasound path

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with Crohn's disease, either:
  * hospitalized for small bowel obstruction, OR,
  * undergoing outpatient start of anti-tumor necrosis factor alpha
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2012-09; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Change in CDAI Score Over 90 days from Hospital Admission | CDAI Score measured over 90 days
  CDAI score will be assessed at 3 time points:
  Hospital Admission Hospital Discharge 90-day follow-up
Shear Wave Velocity | Day 0,3,5,7 of Hospitalization
  Ultrasound shear wave velocity measurements in bowel wall

SECONDARY OUTCOMES:
Need for Re-hospitalization or Surgery within 90 days of discharge | 90 days post discharge
  Telephone follow up with subjects 90 days following index hospitalization to assess need for re-hospitalization or surgery

CONTACTS AND LOCATIONS:
Overall Officials: Ryan W Stidham, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Health System, Ann Arbor, Michigan, United States